CLINICAL TRIAL: NCT03503968
Title: A Phase I/II, Open-Label, Non-Randomized, Multicentre, Dose-Escalation Clinical Trial With Control Group to Evaluate the Safety, Feasibility and Preliminary Efficacy of PRAME TCR Modified T Cells, MDG1011, in Subjects With High Risk Myeloid and Lymphoid Neoplasms
Brief Title: TCR Modified T Cells MDG1011 in High Risk Myeloid and Lymphoid Neoplasms
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The clinical trial is terminated after the completion of phase I without moving to Phase II.
Sponsor: Medigene AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-TCR-001
Record Dates: First submitted 2018-03-21; First posted 2018-04-20 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Safety; Tolerability; Feasibility; Treatment Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase I - 3 disease entities (Experimental): MDG1011 administration of escalating doses
  Interventions: Drug: MDG1011
- Phase II - HLA*02:01 - disease entity 1 (Experimental): MDG1011 administration of Phase II recommended dose
  Interventions: Drug: MDG1011
- Phase II - HLA*other - disease entity 1 (Active Comparator): Investigator Choice therapy
  Interventions: Other: Investigator Choice therapy
- Phase II - HLA*02:01 - disease entity 2 (Experimental): MDG1011 administration of Phase II recommended dose
  Interventions: Drug: MDG1011
- Phase II - HLA*other - disease entity 2 (Active Comparator): Investigator Choice therapy
  Interventions: Other: Investigator Choice therapy

INTERVENTIONS:
Drug: MDG1011 — PRAME-T-Cell Receptor Gene Modified Autologous T Cells
  Arms: Phase I - 3 disease entities; Phase II - HLA*02:01 - disease entity 1; Phase II - HLA*02:01 - disease entity 2
Other: Investigator Choice therapy — Any intervention/therapy chosen by the investigator
  Arms: Phase II - HLA*other - disease entity 1; Phase II - HLA*other - disease entity 2

SUMMARY:
This is a multicentre, non-randomized, open-label, Phase I/II clinical trial of MDG1011, an investigational medicinal product (IMP), consisting of patient-derived autologous T cells, persistently transduced with a Preferentially Expressed Antigen in Melanoma (PRAME)-specific human leukocyte antigen (HLA)-A*02:01-restricted T cell receptor (TCR).

DETAILED DESCRIPTION:
Phase I:

The Phase I dose escalation part will establish the MTD/RP2D in subjects with high risk myeloid and lymphoid neoplasms, a total of 3 disease entities.

Phase I subjects will be enrolled into the following cohorts and treated with a single intravenous (i.v.) infusion of IMP:

* Cohort 1: target dose of 1 x 105 T cells/kg ± 20%
* Cohort 2: target dose of 1 x 106 T cells/kg ± 20%
* Cohort 3: target dose of 5 x 106 T cells/kg ± 20%
* Optional cohort 4: up to 1 x 107 T cells/kg + 20%

Phase II:

The Phase II part consists of two arms, each representing one disease entity. Within each arm, representing a disease entity, subjects will be enrolled in 2 different treatment groups to receive either:

1. IMP in the treatment group (up to 20 subjects who are positive for human leukocyte antigen (HLA)-A*02:01); Or
2. therapy as per Investigator's discretion in the concurrent control (up to 20 subjects who are negative for HLA-A*02:01).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Signed written informed consent prior to any clinical trial-related activities
2. Documented diagnosis with the last disease staging within the last 4 weeks prior to screening
3. Human leukocyte antigen (HLA):

   1. Phase I and Phase II (treatment group): Subjects positive for HLA-A*02:01 according to genotyping results
   2. Phase II (concurrent control group): Subjects negative for HLA-A*02:01 according to genotyping results
4. Age ≥ 18 years
5. Life expectancy of at least 4 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
7. Subjects not planned for allogeneic HSCT (e.g. based on disease characteristics or subject characteristics). Bridging to an allogeneic HSCT will be allowed.
8. Females of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) pregnancy test result before leukapheresis and before administration of lymphodepleting chemotherapy. Females of non-childbearing potential are those who are postmenopausal greater than 2 years or who have had a bilateral tubal ligation or hysterectomy.
9. Females of childbearing potential and males who have partners of childbearing potential must agree to use an effective contraception method during the clinical trial and for 6 months following the last dose of IMP.

Effective birth control includes:

1. intrauterine device plus 1 barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm).

   AML-SPECIFIC INCLUSION CRITERIA:
   1. No Complete remission/response (CR) or Complete remission with incomplete hematologic recovery (CRi) after completion of at least 2 cycles of intensive induction chemotherapy or 1 cycle of intensive induction and consolidation (intermediate or high dose cytarabine) chemotherapy each and/or
   2. No CR or no CRi after completion of at least 1 cycle of intensive induction chemotherapy including at least 5 days of cytarabine 100-200 mg/m^2 continuously or an equivalent regimen with cytarabine with total dose not less than 500 mg/m^2 per cycle and at least 2 days of an anthracycline (e.g. daunorubicine, idarubicin), unable to undergo allogeneic HSCT and/or
   3. Refractory disease (including stable disease [SD], progressive disease [PD]) or relapsed disease after hypomethylating agent therapy (e.g. azacitidine, decitabine) and/or
   4. Any SD, partial response (PR), CRi, CR obtained after re-induction or salvage-therapy and/or
   5. Relapsed AML patients unable to undergo allogeneic HSCT and/or
   6. Relapsed AML after allogeneic HSCT

      1. at least 100 days after transplant
      2. no evidence of active acute or chronic GvHD at enrolment
      3. in case of history of acute (> overall grade 1) or chronic GvHD (moderate/severe) requiring immunosuppression treatment, no immunosuppression within the last 3 months
      4. no immunosuppression (with the exception of low dose steroids <= 10 mg prednisone or equivalent) 4 weeks before enrolment and ongoing and
   7. Myeloid blasts must positively express PRAME

   MDS-SPECIFIC INCLUSION CRITERIA:
   1. IPSS INT-2 or High Grade MDS Excess Blasts-2 (EB-2) not responding to at least 6 courses of azacitidine or 4 courses of decitabine and/or
   2. IPSS INT-1, INT-2 or High Grade MDS with recurrence after initial response and
   3. Blasts must positively express PRAME

   MM-SPECIFIC INCLUSION CRITERIA:
   1. Relapsed and refractory multiple myeloma:

      • Progressive MM, also defined as relapsed disease, defined as:
      1. A 25% increase from baseline in the serum M-protein (absolute increase

         * 0.5 g/dL), urine M-protein (absolute increase > 200 mg/day), and/or the difference between involved and uninvolved free light chain levels (absolute increase ≥ 10 mg/dL).
      2. The presence of definite new bone lesions and/or soft tissue plasmacytomas with a clear increase in the size of existing plasmacytomas, or hypercalcemia, that cannot be attributed to another cause. • Relapsed and refractory MM is defined as disease progression within 60 days of a patient's last treatment where at least a minimal response was achieved. • Primary refractory MM is defined as disease that fails to achieve at least a minimal response with any therapy. and
   2. At least 3 previous therapy lines with at least one proteasome inhibitor and one immunomodulatory derivate (IMiDs). Induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single regimen. and
   3. Myeloma cells must positively express PRAME

      CRITERIA FOR PRE-EMPTIVE LEUKAPHERESIS PROCEDURE

      • subject is positive for HLA-A*02:01 and their blasts/myeloma cells express PRAME

      • subject fulfills at least some inclusion criteria and, based on the judgement of the investigator, have a likelihood of being eligible for IMP administration in the further course of the subjects disease
      * subject does not fulfill any exclusion criterion that would be considered permanent (i.e.

      irreversible organ function impairment) and therefore would certainly preclude the subject from receiving the IMP in the future

      EXCLUSION CRITERIA:

   <!-- -->

   1. Subjects with acute promyelocytic leukemia exhibiting t(15;17)(q22;q12); PML-RARA, or with variant translocations
   2. Pregnant or lactating women
   3. Known positive for HIV, active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
   4. Any clinically significant, advanced or unstable disease or inadequate main organ function that may put the subject at special risk, such as: a. creatinine > 2.0 times the upper normal serum level b. total bilirubin, ALT, AST >3 times the upper normal serum level c. cardiac left ventricular ejection fraction < 40% at rest d. severe restrictive or obstructive lung disease
   5. History of haploidentical allogeneic stem cell transplantation
   6. Subjects both with urinary outflow obstructions and on dialysis or subjects for whom cyclophosphamide is contraindicated for other reasons
   7. Clinical significant and ongoing immune suppression including, but not limited to: immunosuppressive agents such as cyclosporine or corticosteroids (at an equivalent dose of >= 10 mg prednisone per day). Inhaled steroid and physiological replacement for adrenal insufficiency is allowed.
   8. Subjects with currently active autoimmune disease.
   9. Subjects with a history of primary immunodeficiency.
   10. Subjects with a currently active second malignancy other than non- melanoma skin cancers or subjects with history of prior malignancy and previously treated with a curative intent therapy less than 1 year ago
   11. Known or suspected hypersensitivity or intolerance to IMP, cyclophosphamide, fludarabine and/or tocilizumab or to any of the excipients
   12. Participation in any clinical trial < 60 days prior to first IMP administration in case of antibodies and < 14 days for all other IMPs
   13. Vulnerable subjects and/or subjects unwilling or unable to comply with procedures required in this clinical trial protocol

   MM-SPECIFIC EXCLUSION CRITERIA FOR PHASE I AND PHASE II (TREATMENT GROUP):
   1. Prior therapy with IMiDs within 14 days prior to leukapheresis and/or infusion of IMP
   2. Prior therapy with corticosteroids within 7 days prior to leukapheresis or 7 days prior to infusion of IMP

   EXCLUSION CRITERIA FOR TREATMENT WITH IMP IN PHASE I AND PHASE II (TREATMENT GROUP):
   1. Uncontrolled central nervous system (CNS) disease
   2. Uncontrolled infections or uncontrolled disseminated intravascular coagulation; however, if these problems resolve, the start of treatment can be initiated on a delayed schedule
   3. Ongoing 3 grade cardiac, renal, pulmonary, gastrointestinal or hepatic toxicities according to CTCAE v4.03; however, if these problems resolve, the start of treatment can be initiated on a delayed schedule
   4. Evidence of acute or chronic GvHD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Phase I: Adverse Events and Dose Limiting Toxicities (Safety and Tolerability) | 3 months
  Incidence and severity of adverse events according to the NCI CTCAE, v4.03; MTD and/or RP2D of IMP measured by dose-limiting toxicities (DLTs) up to 28 days post infusion
Phase I: maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of MDG101 | 28 days
Phase I: For feasibility: percent of all subjects who receive the planned target dose of MDG1011 | 3 months
Phase II: Adverse Events (Safety) | 3 months
  Incidence and severity of adverse events according to NCI CTCAE, v4.03
Phase II: overall response rate (ORR) | 3 months

SECONDARY OUTCOMES:
Phase I: overall response rate (ORR) | 3, 6 and 12 months
Phase I: time to event and duration of response (DoR) rate | 3, 6 and 12 months
Phase I: time to event and time to progression (TTP) rate | 3, 6 and 12 months
Phase I: time to event and progression-free survival (PFS) rate | 3, 6 and 12 months
Phase I: time to event and overall survival (OS) rate | 3, 6 and 12 months
Phase I: Change in quality of life (QoL) | baseline, 3, 6 and 12 months
  EQ-5D-5L questionaire
Phase I: Change in quality of life (QoL) | baseline, 3, 6 and 12 months
  EORTC-QLQ-C30 [AML/MDS] questionaire
Phase I: Change in quality of life (QoL) | baseline, 3, 6 and 12 months
  EORTC-MY20 [MM] questionaire
Phase I: Correlation of PRAME expression with the antitumor response | 3, 6 and 12 months
Phase II: time to event and duration of response (DoR) rate | 3, 6 and 12 months
Phase II: time to event and time to progression (TTP) rate | 3, 6 and 12 months
Phase II: time to event and progression-free survival (PFS) rate | 3, 6 and 12 months
Phase II: time to event and overall survival (OS) rate | 3, 6 and 12 months
Phase II: changes in quality of life (QoL) | baseline, 3, 6 and 12 months
  EQ-5D-5L questionaire
Phase II: changes in quality of life (QoL) | baseline, 3, 6 and 12 months
  EORTC-QLQ-C30 [AML/MDS] questionaire
Phase II: changes in quality of life (QoL) | baseline, 3, 6 and 12 months
  EORTC-MY20 [MM] questionaire
Phase II: For feasibility, the percent of all subjects who receive the RP2D of MDG1011 | 3 months
Phase II: correlation of PRAME expression with the antitumor response | 3, 6 and 12 months
Phase I: Adverse Events (safety) | 6 and 12 months
  Incidence and severity of adverse events according to NCI CTCAE, v4.03
Phase II: Adverse Events (safety) | 6 and 12 months
  Incidence and severity of adverse events according to NCI CTCAE, v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Simone Thomas, PD Dr. med., Principal Investigator — University Hospital Regensburg
Locations (9):
- Germany (9):
  - University Hospital Dresden, Dresden
  - University Hospital Erlangen, Erlangen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Leipzig, Leipzig
  - University Hospital Mainz, Mainz
  - University Hospital Regensburg, Regensburg
  - University Hospital Wuerzburg, Würzburg

REFERENCES:
- [Derived] Burdek M, Prinz PU, Mutze K, Tippmer S, Geiger C, Longinotti G, Schendel DJ. Characterization of a 3S PRAME VLD-Specific T Cell Receptor and Its Use in Investigational Medicinal Products for TCR-T Therapy of Patients with Myeloid Malignancies. Cancers (Basel). 2025 Jan 13;17(2):242. doi: 10.3390/cancers17020242. PMID 39858024